CLINICAL TRIAL: NCT04211441
Title: An Initial Assessment of Safety and Performance of the Sphere-9™ Catheter and System for Mapping and Ablation of Atrial and Ventricular Arrhythmias
Brief Title: Assessment of the Sphere-9™ Catheter and Affera Mapping and Ablation System for Treatment of Atrial and Ventricular Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00001-E
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Ventricular Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects who are treated with the Sphere-9™ Catheter (Experimental)
  Interventions: Device: Catheter mapping and ablation with the Sphere-9 Catheter and Affera Mapping and Ablation System

INTERVENTIONS:
Device: Catheter mapping and ablation with the Sphere-9 Catheter and Affera Mapping and Ablation System — Catheter mapping and ablation with the Sphere-9 Catheter and Affera Mapping and Ablation System

SUMMARY:
A prospective, single-arm, multi-center, safety and performance assessment of the Sphere-9™ Catheter and the Affera Mapping and RF Ablation System to treat Atrial Arrhythmias

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 75 years.
2. Suitable candidate for catheter non-emergent mapping and ablation of cardiac arrhythmia as follows:

   • Atrial Flutter (AFL) defined as

   o At least one episode of typical (clockwise or counterclockwise) atrial flutter documented by EKG, 12 lead EKG, Holter or transtelephonic monitor, telemetry strip, or implanted device within 6 months prior to enrollment.

   OR

   • Atrial Fibrillation (AF) defined as
   * History of symptomatic paroxysmal and/or persistent atrial fibrillation within the past year documented by EKG AND
   * Failure of at least one class I-IV drug as evidenced by recurrent symptomatic AF, or intolerable to AAD.
3. Subject is able and willing to give informed consent.
4. Subject is able and willing, and has ample means to comply with all pre-, post- and follow-up testing requirements.

Exclusion Criteria:

1. Documented thrombus or another abnormality which precludes catheter introduction.
2. Documented ejection fraction (EF) < 40% for AF and AFL, and EF < 15% for VT.
3. Contraindication to anticoagulation therapy (heparin, warfarin, or novel oral anticoagulant [NOAC]).
4. Unstable angina or ongoing myocardial ischemia.
5. Myocardial infarction, unstable angina, cardiac surgery or coronary intervention within 3 months of enrollment.
6. Congenital heart disease where the underlying abnormality increases the risk of the ablation.
7. Pulmonary hypertension (mean pulmonary artery pressure [mPAP] > 50 mmHg)
8. Enrollment in any other ongoing study protocol that would interfere with this study.
9. Documented severely impaired kidney function defined as Cockcroft-Gault Glomerular Filtration Rate (GFR) < 29ml/min.
10. Active gastrointestinal (GI) bleeding.
11. Active infection or sepsis.
12. Short life expectancy (< 1 year) due to illness such as cancer, pulmonary, hepatic or renal disease.
13. Significant anemia (defined as hemoglobin < 8.0 gr/dL).
14. Severe uncontrolled systemic hypertension with systolic blood pressure (SBP) > 200 mm Hg within last 30 days.
15. Severe bleeding, clotting or thrombotic disorder.
16. Uncontrolled diabetes.
17. Women who are pregnant or are not willing to use contraception for the duration of the study.
18. Severe chronic obstructive pulmonary disease (COPD; identified by a forced expiratory volume [FEV1] <1)
19. Prior stroke or TIA within the last 6 months.
20. Prior atrial septal defect (ASD) or patent foramen ovale (PFO) closure with a device using a transcatheter percutaneous approach.
21. Hypertrophic cardiomyopathy defined as left ventricular (LV) septal wall thickness >1.5cm.
22. Any other condition that, in the opinion of the investigator, poses a significant hazard to the subject if an ablation procedure was performed.

    Additional exclusion criteria for AF patients only:
23. Left atrial diameter of >55 mm (parasternal view).
24. Prior ablation or surgery for atrial fibrillation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neužil, MD. PhD., Principal Investigator — Homolka Hospital, Prague; Petr Peichl, MD. PhD., Principal Investigator — Institute Klinicke a Experimentalni Mediciny
Locations (2):
- Czechia (2):
  - Homolka Hospital, Prague
  - Institute Klinicke a Experimentalni Mediciny, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkagan M, Leshem E, Rottmann M, Sroubek J, Shapira-Daniels A, Anter E. Expandable Lattice Electrode Ablation Catheter: A Novel Radiofrequency Platform Allowing High Current at Low Density for Rapid, Titratable, and Durable Lesions. Circ Arrhythm Electrophysiol. 2019 Apr;12(4):e007090. doi: 10.1161/CIRCEP.118.007090. PMID 30943762
- [Background] Kitamura T, Hocini M, Bourier F, Martin R, Takigawa M, Frontera A, Thompson N, Cheniti G, Vlachos K, Martin CA, Lam A, Duchateau J, Pambrun T, Denis A, Sacher F, Derval N, Cochet H, Haissaguerre M, Jais P. Larger and deeper ventricular lesions using a novel expandable spherical monopolar irrigated radiofrequency ablation catheter. J Cardiovasc Electrophysiol. 2019 Sep;30(9):1644-1651. doi: 10.1111/jce.14089. Epub 2019 Aug 1. PMID 31347223

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 subjects were enrolled in the study. Of these, five were excluded or withdrew prior to treatment with the study devices. 69 patients underwent the procedure.
Groups:
- Sphere-9™ Catheter: Catheter mapping and ablation with the Sphere-9 Catheter and Affera Mapping and Ablation System: Catheter mapping and ablation with the Sphere-9 Catheter and Affera Mapping and Ablation System
Period: Overall Study
Arm/Group | Sphere-9™ Catheter
Started | 74
Completed | 61
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Baseline subject demographics for all subjects treated with the investigational device.
Arm/Group | Sphere-9™ Catheter
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Primary Safety Event
Description: The primary safety outcome is the rate of the following serious adverse events (SAEs) occurring starting Day 0 and extending through the Day 10 post-treatment assessment: transient ischemic attack; cerebrovascular accident; major bleeding; cardiac tamponade; pulmonary vein stenosis; severe pericarditis requiring extended hospitalization; myocardial infarction; diaphragmatic paralysis; atrio-esophageal fistula (through the Day 90 assessment) ; valvular damage; phrenic nerve palsy; intra-procedural device complications requiring open chest or heart surgery; vascular complications requiring surgical intervention; and death.
Time Frame: 90 days
Population: Subjects who underwent a procedure with the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9™ Catheter
Number analyzed (Participants) | 69
Participants | 2

2. Primary Outcome: Number of Positive (Affirmative) Product Performance Responses
Description: The primary acute product performance outcome is determined during the procedure and is defined as the following:
  * Catheter handling sufficient to reach reasonable intended targets, as determined by the physician:
    * catheter delivery to the desired cardiac chambers
    * manipulation of catheter
    * completion of mapping procedure
    * safe removal of catheter from the subject
  * 3D electro-anatomical map creation and utility sufficient to aid diagnosis
  * Generation of acceptable acute therapeutic RF lesions
Time Frame: Index ablation procedure
Population: All ablation procedures using the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9™ Catheter
Number analyzed (Participants) | 69
Participants | 69

3. Secondary Outcome: Percentage of Subjects Free From Documented Recurrence
Description: A secondary product effectiveness outcome is freedom from documented recurrence of the treated arrhythmia through the Day 365 post-treatment follow-up visit. In AF subjects, this includes freedom from documented AF, atrial tachycardia (AT), or AFL.
Time Frame: 12 months
Population: Subjects treated for AF
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9™ Catheter
Number analyzed (Participants) | 20
Participants | 19

4. Secondary Outcome: Number of Patients With Durable Ablation Lesions at Remapping Procedure
Description: * In AF subjects that are remapped, the number of pulmonary veins that remain isolated and the number of patients with all pulmonary veins isolated will be determined.
  * In all subjects that are remapped, the number of previously confirmed lines of block remaining isolated will be determined.
Time Frame: 3 months
Population: Subset of subjects treated for AF underwent a remapping procedure to assess durability
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9™ Catheter
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Sphere-9™ Catheter
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 5/69
Other Adverse Events (participants affected / at risk) | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sphere-9™ Catheter (N=69)
Pericarditis (Cardiac disorders) | 1 (1)
Esophogeal thermal injury (Skin and subcutaneous tissue disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Diaphragmatic paralysis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT04211441/Prot_SAP_000.pdf